CLINICAL TRIAL: NCT01840878
Title: Accuracy of Actigraph Measured Sleep Compared to Polysomnography During Acute Uncomplicated Diverticulitis
Brief Title: Validation of Actigraph Measured Sleep During Acute Diverticulitis
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Ismail Gögenür, Senior resident and D.Sc., Herlev Hospital
Other Study IDs: CHU-2
Record Dates: First submitted 2013-04-13; First posted 2013-04-26 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Acute Diverticulitis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute Diverticulitis: CT-verified acute uncomplicated diverticulitis managed by antibiotics

SUMMARY:
The purpose of this study is to investigate the accuracy of actigraph measured sleep compared to the golden standard (polysomnography) during Acute uncomplicated diverticulitis. Our hypothesis is the actigraph is accurate for sleep-monitoring for this group of patients

DETAILED DESCRIPTION:
The actigraph has been proven to measured sleep data with an accuracy about 80% (compared with Polysomnography) in patients who have undergone surgery.

But this accuracy has not been validated in relation to none surgical inflammatory diseases. This study will investigate the accuracy of actigraph measured sleep in diverticulitis patients.

Following methods will be applied

Device: Wrist-Actigraph - Octagonal Basic Motionlogger, Ambulatory monitoring Inc, New York, USA

Other: Sleep-diary

Device: Polysomnograph - Embla Titanium (Natus Medical Incorporated, USA)

ELIGIBILITY:
Inclusion Criteria:

* CT-verified diverticulitis patients managed by antibiotic treatment at Herlev Hospital
* Pain and fever occurred less than 72 hours prior to the admission
* ASA (American Society of Anesthesiologists) score I to III

Exclusion Criteria:

* Surgical intervention needed
* Complicated diverticulitis
* Complications in relation to diverticulitis
* Pain and fever occurred more than 72 hours prior to the admission
* In anticoagulant treatment and heart rate control treatment
* Known Autoimmune disease
* Known medically treated sleep-disorder (insomnia, restless legs etc.) and sleep apnea
* Shift-work or jetlag
* Daily use of opioid, psychopharmaca, opioids or anxiolytics (including Hypnotics)
* Known psychiatry conditions in treatment with psychopharmaca
* Daily alcohol intake of more than 5 units or drug abuse
* Missing written consent
* Diabetes Mellitus
* Predicted bad compliance
* Pregnant or breast-feeding
* Urine or fecal incontinence
* Severe kidney disease
* Current cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 16 x Acute uncomplicated diverticulitis (Hansen and stock stage 1) patients aged 18-75 years managed by antibiotic treatment at Herlev Hospital.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Changes in Sleep data during acute uncomplicated diverticulitis (1-5th days following the admission) from baseline at remission (5th-30th days) | 1st-30th days following the admission
  Sleep measured by Actigraphy (total minutes asleep, sleep effectiveness, sleep latency, awakenings). A wrist actigraph wil be worn from 1st day of the admission and taken off on the 31st day.
Changes in Circadian rhythm during acute uncomplicated diverticulitis (1-5th days following the admission) from baseline at remission (5th-30th days) | 1st-30th days following the admission
  Circadian rhythm measured by Actigraphy. A wrist actigraph wil be worn from 1st day of the admission and taken off on the 31st day.
Accuracy of actigraphy measured sleep data in compare to Polysomnography both in inflammatory condition and in remission condition | 1st, 2nd and 30th days following the admission
  Sleep data measured by Actigraphy (total minutes asleep, sleep effectiveness, sleep latency, awakenings) are to validate with the PSG-measured data

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, M.D., Principal Investigator — University of Copenhagen, Herlev Hospital
Locations (1):
- Department D, Herlev Hospital, Herlev, Copenhagen, Denmark